CLINICAL TRIAL: NCT04605510
Title: Acute Effect of Passive Joint Mobilization on Joint Motion And Pain Perception in Non-Specific Neck Pain
Brief Title: Acute Effect of Passive Joint Mobilization in Non-Specific Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mücahit ÖZTOP (Other)
Collaborators: Pamukkale University (Other)
Responsible Party: Sponsor-Investigator, Mücahit ÖZTOP, Research Assistant, Pamukkale University
Organization: Pamukkale University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 60116787-020/46072
Record Dates: First submitted 2020-10-22; First posted 2020-10-28 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Neck Pain
Keywords: non-specific neck pain; passive joint mobilization; blood markers; neck range of motion
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: This study includes two groups. Intervention group including women with non-specific neck pain will applied cervical passive joint mobilization and assessment protocol. Control group including healthy women without pain will applied only assessment protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): 24 female participants with non-specific neck pain included in the mobilization group will undergo detailed manual cervical examination. In the evaluation, the most painful segment with dysfunction will be selected and mobilization application and algometric measurements will be performed on this segment. Grade 3 Central Posterior-Anterior (CPA) passive joint mobilization with Maitland method will be applied in 3 sets, 30 seconds, to the segment with the detected dysfunction.
  Interventions: Other: Passive Cervical Joint Mobilization
- Healthy Control Group (No Intervention): Healthy volunteer participants included in the control group will only be applied an evaluation protocol and blood samples will be taken without any application.

INTERVENTIONS:
Other: Passive Cervical Joint Mobilization — It will be applied to the cervical spine, whose dysfunction is detected as a result of the evaluation. The participant will be in the prone position and Grade 3 Central Posterior-Anterior (CPA) passive joint mobilization with Maitland method will be applied for 3 sets, 30 seconds, to the segment to be treated.
  Other Names: Maitland Mobilization
  Arms: Intervention Group

SUMMARY:
Aim of present study is investigating the acute effects of passive joint mobilization on pain perception and range of motion. Study protocol includes passive joint mobilization application to study group with neck pain and blood sample collection of study and healthy control group.

DETAILED DESCRIPTION:
Our purpose of planning this study is to examine the acute effect of passive joint mobilization application on pain perception and range of motion in women with non-specific neck pain.

The hypotheses we will test for this purpose;

H1- Passive joint mobilization application increases the range of motion of the cervical joint in women with non-specific neck pain.

H2- Passive joint mobilization application increases the pressure pain threshold in women with non-specific neck pain.

H3- Passive joint mobilization increases serum Orexin A and Neurotensin levels in women with non-specific neck pain.

ELIGIBILITY:
Inclusion Criteria:

For Intervention Group;

* Having neck pain lasting more than 30 days and being diagnosed with non-specific neck pain
* Having obtained 14/50 points and above in Neck Disability Index
* Expressing neck pain at least 34/100 points and above on a Visual Analog Scale
* Being 20-45 years old and female

For Healthy Control Group;

- Healthy volunteers without a chronic illness and musculoskeletal pain

Exclusion Criteria:

* Congenital anomalies
* Previously diagnosed orthopedic diseases related to the spine
* Pregnancy and having just given birth
* Within the last 3 months; use of corticosteroids, cytotoxic drugs, or immunosuppressants
* Liver or kidney failure
* Acute or chronic infections (including HIV)
* Serious pathologies (such as cancer, spondylolisthesis, rheumatoid arthritis or ankylosing spondylitis)
* Symptoms of cervical spinal stenosis (such as incoordination of hands, arms and legs, bowel and bladder incontinence)
* Radix compression (such as sensory changes, muscle weakness or decreased reflexes)
* Whiplash or a history of cervical surgery

Ages: 24 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2022-05-23 (Actual)

PRIMARY OUTCOMES:
Cervical Range of Motion | Cervical Range of Motion assessment will take maximum of 5 minutes.
  Cervical Range of Motion will be assessed by Baselşne Bubble Inclinometer as degree of flexion-extension, rotation and lateral flexion and will be recorded.
Pain Pressure Threshold | Pain Pressure Threshold assessment will take maximum of 5 minutes.
  Pressure Pain Threshold will be measured with the JTech Commander Algometer at the level of the right and left zygapophyseal joint of the dysfunctional cervical segment detected during physical examination. During the evaluation, the participants will be asked to lie in a prone position. By placing the probe of the algometer vertically on the skin, the pressure applied will be gradually increased and the participant will be asked to report at the first moment of pain. The measurement will be made once and the result will be recorded in kilograms.
Neuropeptide Measurement | Blood Sample Collection for Neuropeptide Measurement will take maximum of 5 minutes.
  Neuropeptide Measurement will be performed as a result of evaluating the blood samples taken from the participants with the appropriate ELISA kits. Orexin A and Neurotensin levels are planned to be evaluated with Human Orexin A (Competitive EIA) ELISA Kit and Human NTS / NT / Neurotensin (Competitive EIA) ELISA Kit which are specific for these neuropeptides.

SECONDARY OUTCOMES:
Pain Intensity Measurement | Pain Intensity Measurement will take maximum of 1 minute.
  Pain intensity will be evaluated with the Visual Analogue Scale. The Visual Analogue Scale is a horizontal scale in the range of 0-100 mm, where 0 is the lowest pain and 100 the highest pain. The patient will be asked to mark the pain felt in the neck area on this line and the point marked will be measured with a ruler and recorded in mm.
Neck Disability | Neck Disability measurement will take maximum of 1 minute.
  Neck Disability will be measured by Neck Disability Index. The Neck Disability Index is a frequently used scale to evaluate the level of disability due to neck pain. It consists of 10 items and 6 options under each item. Options are scored between 0-5 points. An increasing score indicates a higher level of disability. The minimum score that can be obtained from the scale is 0, and the highest score is 50. 14 points are used as cut-off points for the minimal level of disability.

CONTACTS AND LOCATIONS:
Overall Officials: Nesrin YAĞCI, Professor, Study Director — Pamukkale University School of Physical Therapy and Rehabilitation
Locations (1):
- Pamukkale University School of Physical Therapy and Rehabilitation, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Plaza-Manzano G, Molina-Ortega F, Lomas-Vega R, Martinez-Amat A, Achalandabaso A, Hita-Contreras F. Changes in biochemical markers of pain perception and stress response after spinal manipulation. J Orthop Sports Phys Ther. 2014 Apr;44(4):231-9. doi: 10.2519/jospt.2014.4996. Epub 2014 Jan 22. PMID 24450367
- [Background] Molina-Ortega F, Lomas-Vega R, Hita-Contreras F, Plaza Manzano G, Achalandabaso A, Ramos-Morcillo AJ, Martinez-Amat A. Immediate effects of spinal manipulation on nitric oxide, substance P and pain perception. Man Ther. 2014 Oct;19(5):411-7. doi: 10.1016/j.math.2014.02.007. Epub 2014 Mar 5. PMID 24674816
- [Background] Lohman EB, Pacheco GR, Gharibvand L, Daher N, Devore K, Bains G, AlAmeri M, Berk LS. The immediate effects of cervical spine manipulation on pain and biochemical markers in females with acute non-specific mechanical neck pain: a randomized clinical trial. J Man Manip Ther. 2019 Sep;27(4):186-196. doi: 10.1080/10669817.2018.1553696. Epub 2018 Dec 11. PMID 30935335
- [Background] Maitland GD. Maitland's Vertebral Manipulation. Seventh Ed. (Hengeveld E, Banks K, eds.). Edinburgh; New York: Churchill Livingstone; 2013. https://www.elsevier.com/books/maitlands-vertebral-manipulation/hengeveld/978-0-7020-4066-5.